CLINICAL TRIAL: NCT06589505
Title: A Multicenter, Randomized, Double-blind, Parallel-group Comparative Study to Assess Efficacy and Safety of Software as a Medical Device in Patients With Post-Traumatic Stress Disorder (PTSD)
Brief Title: Software as a Medical Device for the Treatment of Patients With PTSD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Otsuka Medical Devices Co., Ltd. Japan (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 380-102-0001
Record Dates: First submitted 2024-08-22; First posted 2024-09-19 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Post-Traumatic Stress Disorder, PTSD
MeSH Terms: conditions — Combat Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Software as a Medical Device1 (Experimental)
  Interventions: Device: Software as a Medical Device
- The Software as a Medical Device2 (Other)
  Interventions: Device: Software as a Medical Device

INTERVENTIONS:
Device: Software as a Medical Device — The subject will undergo treatment using the Software as a Medical Device

SUMMARY:
To evaluate the efficacy and safety of Software as a Medical Device in patients with Post-Traumatic Stress Disorder (PTSD)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD according to the DSM-5
* Subjects who are within 1 to 20 years since index trauma

Exclusion Criteria:

* Subjects diagnosed with schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, bipolar I disorder, autism spectrum disorder, or intellectual disability based on DSM-5.
* Subjects diagnosed with any mood disorder and anxiety disorder according to DSM-5 that is the primary focus of treatment in the last 6 months prior to screening, as per the clinical judgement of the investigator
* Subjects who have completed two or more full courses of trauma-focused therapy in the past

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 | baseline and after intervention (up to 21 weeks)
  The primary objective of this study is to assess the change from baseline of the Clinician Administered PTSD Scale (CAPS - 5) score.
  Scores range from 0 - 80, with higher scores indicating increased PTSD symptom severity.

CONTACTS AND LOCATIONS:
Locations (35):
- Japan (35):
  - Yamanashi Prefectural Kita Hospital, Yamanashi, Hokkaido
  - Heart Care Clinic Omachi, Akita
  - Aburayama Hospital, Fukuoka
  - Ai Sakura Clinic, Fukuoka
  - Hatakeyama Clinic, Fukuoka
  - Hiro Mental Clinic, Fukuoka
  - Hirota Clinic, Fukuoka
  - Kurume University Hospital, Fukuoka
  - Medical corporation Shinseikai Kaku Mental Clinic, Fukuoka
  - Mental Clinic Sakurazaka, Fukuoka
  - Nishie Kokorono Clinic, Fukuoka
  - Uematsu Mental Clinic, Fukuoka
  - PTSD Care Matsumoto Mental Clinic, Gunma
  - Goryokai Hospital, Hokkaido
  - Sakamoto Misako Mental Clinic, Hyōgo
  - Takahashi Psychiatric Clinic, Hyōgo
  - Tsukuba Psychosomatics Clinic, Ibaraki
  - Musashikosugi J Kokorono Clinic, Kanagawa
  - Niki Hearty Hospital, Kumamoto
  - Arata Clinic, Nagasaki
  - Okayama Psychiatric Medical Center, Okayama
  - Barclay Imuro Mental Clinic, Okinawa
  - Medical Corporation Mikokorokai Shimizu Clinic, Osaka
  - Sho Midori Hospital, Saitama
  - Ai Mental Clinic, Tochigi
  - i Kokoro Clinic Nihonbashi, Tokyo
  - Iidabashi Mental Clinic, Tokyo
  - Ikebukuro Olive Mental Clinic, Tokyo
  - Kitaikebukuro Kokoro No Clinic, Tokyo
  - Maynds Tower Mental Clinic, Tokyo
  - Monzennakacho Mental Clinic, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - Sakurazaka Clinic SophyAnce, Tokyo
  - Sangenjaya Nakamura Mental Clinic, Tokyo
  - Wakamatsucho Kokoro to Hifu Clinic, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided